CLINICAL TRIAL: NCT03747484
Title: ATTAC-MCC: Phase I/II Study of Autologous CD8+ and CD4+ Transgenic T Cells Expressing High Affinity MCPyV-specific TCRs Combined With Avelumab and Class I MHC-upregulation in Patients With Metastatic MCC Refractory to PD-1 Axis Blockade
Brief Title: Gene-Modified Immune Cells (FH-MCVA2TCR) in Treating Patients With Metastatic or Unresectable Merkel Cell Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Affini-T Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Joshua Veatch, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RG1003611; NCI-2018-02483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9845 (Registry Identifier: Fred Hutch/University of Washington Cancer Consortium); ATTAC-MCC (Other: Collaborator); P01CA225517 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Other Skin
Keywords: Clinical Stage III Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Merkel Cell Carcinoma AJCC v8; Pathologic Stage III Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIA Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIB Merkel Cell Carcinoma AJCC v8; Pathologic Stage IV Merkel Cell Carcinoma AJCC v8; Merkel cell carcinoma, metastatic; Merkel cell carcinoma, unresectable; Metastatic Merkel Cell Carcinoma; Unresectable Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neoplasm Metastasis | interventions — avelumab; B7-H1 Antigen; pembrolizumab; interferon gamma-1b; Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (TCR-T cells, avelumab or pembrolizumab) (Experimental): Approximated 5-7 days prior to receiving FH-MCVA2TCR T-cells, patients receive interferon gamma administered at the FDA-approved dosing of 50mcg/m2, 3 times weekly for a total of 4 weeks. Patients receive FH-MCVA2TCR T-cells IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells.
  Interventions: Biological: Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR; Drug: Avelumab; Biological: Pembrolizumab; Biological: Interferon Gamma-1b
- Treatment 2 (TCR-T cells, avelumab or pembrolizumab) (Experimental): Approximated 5-7 days prior to receiving FH-MCVA2TCR T-cells, patients receive interferon gamma administered at the FDA-approved dosing of 50mcg/m2, 3 times weekly for a total of 4 weeks. Patients receive FH-MCVA2TCR T-cells IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells.
  Interventions: Biological: Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR; Drug: Avelumab; Biological: Pembrolizumab; Biological: Interferon Gamma-1b

INTERVENTIONS:
Biological: Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR — Given IV
  Other Names: Autologous CD8+ and CD4+ T-cells transduced with TCR A2-MCC1; FH-MCVA2TCR; FH-MCVA2TCR Autologous CD8+ and CD4+ T-cells Transduced with TCR A2-MCC1
Drug: Avelumab — Given IV
  Other Names: 1537032-82-8; Bavencio; Immunoglobulin G1-lambda1; Anti-(Homo sapiens CD274 (Programmed Death Ligand 1, PDL1, pd-l1, B7 Homolog 1, B7H1)); Homo sapiens Monoclonal Antibody; MSB-0010718C; MSB0010718C
Biological: Pembrolizumab — Given IV
  Other Names: Anti-(Human Programmed Cell Death 1); Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Interferon Gamma-1b — Given SC
  Other Names: 98059-61-1; Actimmune; gamma Interferon 1B; IFN-g-1b; IFN-gamma 1b; Recombinant Interferon Gamma-1b

SUMMARY:
This phase I/II trial studies the side effects of gene-modified immune cells (FH-MCVA2TCR) and to see how well they work in treating patients with Merkel cell cancer that has spread to other parts of the body (metastatic) or that cannot be removed by surgery (unresectable). Placing a gene that has been created in the laboratory into immune cells may improve the body's ability to fight Merkel cell cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a dose escalation study of FH-MCVA2TCR autologous T-cells.

Patients receive interferon gamma-1b subcutaneously (SC) on study. Patients receive FH-MCVA2TCR T-cells intravenously (IV) over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells.

After completion of study treatment, patients are followed up periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* EVALUATION: Metastatic or unresectable Merkel cell polyomavirus (MCPyV)-associated Merkel cell carcinoma (VP-MCC) that has progressed on or after prior treatment with a PD-1 axis immune checkpoint inhibitor.
* EVALUATION: Individuals that may be consented to undergo evaluation to determine potential eligibility must have a history of metastatic or unresectable Merkel cell carcinoma (MCC) (as documented by medical record).
* EVALUATION: Be 18 years of age or older.
* EVALUATION: Be capable of understanding and providing informed consent.
* Participants must have metastatic or unresectable, histologically confirmed virus-positive MCC. Confirmation of diagnosis must be or have been performed by internal pathology review of initial or subsequent biopsy or other pathologic material at Fred Hutch/Seattle Cancer Care Alliance (SCCA).
* Approximately 80% of MCCs are caused by Merkel cell polyomavirus (MCPyV) T Antigens and the treatment is expected to only be effective in this population. Merkel cell polyomavirus positivity may be established through one of two means: positive Merkel cell polyomavirus T antigen serology (preferred) or immunohistochemistry of a primary or metastatic MCC tumor lesion (if T antigen seronegative).
* MCPyV T Antigen serology will be performed with the anti-Merkel cell panel (AMERK) assay run through the University of Washington Medical Center Laboratory Medicine Clinical Immunology Laboratory. Positivity will be defined as a Merkel oncoprotein antibody titer (MSCTT) of >= 75 standard titer units (STU) at any time point from initial diagnosis onward. Patients with negative T antigen serology but MCPyV positive tumor by other methodologies will be considered for additional MCPyV testing as clinically appropriate, as the T antigen serology assays are highly specific but incompletely sensitive for MCPyV status. In this case, immunohistochemistry of any tumor lesion will be performed with the CM2B4 Merkel cell polyomavirus T antigen antibody. Expression of MCPyV in at least 10% of tumor cells will be considered positive. CM2B4 staining performed at any point clinically and at any clinical laboratory may be accepted. However, if CM2B4 staining has not been previously performed by a clinical pathology laboratory as part of MCC diagnostic workup, it will be performed in a clinical diagnostic pathology laboratory at University of Washington (UW)/Fred Hutchinson Cancer Research Center (FHCRC)/SCCA as per standard staining protocols. Persons are not required to have both CM2B4 positivity and seropositivity; either will be acceptable confirmation of viral status and if one negative and the other positive the patient will remain eligible provided other criteria are met.
* Patients must have been previously treated with at least one dose of a PD-1 axis inhibitor (e.g. PD-1 or PD-L1 inhibiting monoclonal antibody such as pembrolizumab, nivolumab, avelumab, atezolizumab, durvalumab), developed progression of their MCC tumor on or after treatment, or have biopsy confirmed residual disease following treatment. At least four weeks must have passed between the administration of the first dose of PD-1 axis inhibitor and determination of progression or residual disease. If there is significant clinical concern for pseudoprogression (i.e. progression developed rapidly after checkpoint inhibitor therapy), biopsy must be performed to demonstrate true progression. Patients may have received 1 or more prior systemic regimens for MCC. There is no upper limit on prior regimens. Patients may have received prior anti-PD-1/anti-PD-L1 in the neoadjuvant or adjuvant setting. Patients are also eligible if they have a contraindication to PD-1/PD-L1 axis blockade such as a history of an autoimmune disease.
* Participants must be HLA-A*02:01 in order for infused transgenic T cells to recognize antigen-MHC complexes. HLA typing for HLA-A2 should be determined through molecular approaches at a clinical laboratory licensed for HLA testing.
* Life expectancy must be anticipated to be > 3 months at trial entry.
* 18 years of age or older. Fewer than 0.5% of MCC occur in individuals aged 30 years or younger, thus the protocol includes only adult patients.
* Capable of understanding and providing a written informed consent.
* If fertile, willingness to comply with reproductive requirements.
* Karnofsky performance status of >= 60%.
* Should there be no tumor tissue that is accessible for biopsy, patients will still be considered for participation, at discretion of the investigator. Similarly, should an investigator determine that a biopsy cannot be performed safely for clinical reasons biopsies may be cancelled or retimed.
* At least 3 weeks must have passed since any: immunotherapy (for example, T-cell infusions, immunomodulatory agents, interleukins, MCC vaccines, intravenous immunoglobulin, expanded polyclonal tumor infiltrating lymphocyte [TIL] or lymphokine-activated killer cell [LAK] therapy), natural killer (NK) therapy, small molecule or chemotherapy cancer treatment, other investigational agents or other systemic agents that target MCC. There is no washout period for radiation.
* Serum creatinine < 2.5 or estimated glomerular filtration rate (eGFR) > 30.
* Total bilirubin (tBili) < 3.0. Patients with suspected Gilbert syndrome may be included if Tbili > 3 but no other evidence of hepatic dysfunction.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN).
* =< grade 1 dyspnea.
* Oxygen saturation (SaO2) >= 92% on ambient air.
* If pulmonary function tests (PFTs) are performed based on the clinical judgment of the treating physician, patients with forced expiratory volume in one second (FEV1) >= 50% of predicted and diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) of >= 40% of predicted will be eligible.
* Patients 60 years of age or older are required to have left ventricular ejection fraction (LVEF) evaluation performed within 1 year prior to study treatment. LVEF may be established with echocardiogram or multigated acquisition (MUGA) scan, and must be >= 35%. Cardiac evaluation for other patients is at the discretion of the treating physician.
* Absolute neutrophil count (ANC) > 1000 cells/mm^3.
* Absolute lymphocyte count (ALC) > 200 cells/mm^3.
* Hematocrit (HCT) > 30%.
* Platelet count > 50K.

Exclusion Criteria:

* Active autoimmune disease requiring immunosuppressive therapy is excluded unless discussed with the principal investigator (PI). Patients with a history of autoimmune disease that was a contra-indication to PD-1 axis blockade treatment will be eligible, but will not receive PD-1 axis blockade treatment on trial.
* Kidney transplant will be considered on a case by case basis requiring discussion with PI. If kidney transplant, patient must have dialysis access, dialysis plan, supportive nephrologist, willingness to stop transplant immunosuppression, and express understanding that rejection is likely. Dialysis or costs related to transplant kidney will not be supported by the study. Participants having had any other solid organ transplants will be excluded, as will those with a history of allogeneic stem cell transplant.
* Corticosteroid therapy at a dose equivalent of > 10 mg prednisone per day.
* Concurrent use of other investigational agents or MCC directed therapies.
* Any medical or psychological condition other than Merkel cell carcinoma that would significantly increase the risk of harm to a subject or interfere with the interpretation of trial endpoints.
* Active uncontrolled infection. Human immunodeficiency virus (HIV) positive participants on highly active antiretroviral therapy (HAART) with a CD4 count > 500 cells/mm^3 are considered controlled, as are individuals with a history of hepatitis C who have successfully completed antiviral therapy with an undetectable viral load, and those with hepatitis B who have hepatitis well controlled on medication.
* Uncontrolled concurrent illness. Participants may not have uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Untreated brain metastases. Participants with small asymptomatic brain metastases (< 1 cm) or those with brain metastases previously treated with surgery or radiotherapy will be considered for inclusion at discretion of principal investigator, so long as other eligibility criteria are met.
* Grade 3 or higher immune related adverse event (iRAE) to any prior PD-1 axis blocking agent. iRAEs are persistent T cell mediated inflammatory syndromes caused by PD-1 or PD-L1 inhibitors including colitis, nephritis, pneumonitis, myositis, hepatitis, encephalitis.
* Participants receiving treatment for prior immune-related adverse event (iRAE) are excluded, with exception of hormone supplementation or corticosteroid therapy at equivalent of up to 10 mg prednisone per day, unless otherwise approved by PI.
* Study participants must not have significant active underlying neurologic disease, unless approved by PI. Mild neuropathy related to diabetes or prior chemotherapy is acceptable.
* Other medical, social, or psychiatric factor that interferes with medical appropriateness and/or ability to comply with study, as determined by PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Veatch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Radiation + One Infusion at DL1: Following treatment with single fraction radiation to a single lesion, patients receive FH-MCVA2TCR T-cells IV at Dose Level 1 over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
  Pembrolizumab: Given IV
- Cohort 2 - Radiation + One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients receive FH-MCVA2TCR T-cells IV at Dose Level 2 over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
  Pembrolizumab: Given IV
- Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients received FH-MCVA2TCR T-cells at Dose Level 1 IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also received standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells at Dose Level 2.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
  Pembrolizumab: Given IV
- Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2: Following lymphodepleting chemotherapy with fludarabine and cyclophosphamide, patients received FH-MCVA2TCR T-cells at Dose Level 1 IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also received standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells at Dose Level 2.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
  Pembrolizumab: Given IV
- Cohort 5 - Interferon Gamma + One Infusion at DL1: Following treatment with interferon gamma given subcutaneously three times per week for 4 weeks starting 5-7 days before T cell infusion, patients receive FH-MCVA2TCR T-cells IV at Dose Level 1 over 60-120 minutes. Beginning14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
  Pembrolizumab: Given IV
  Interferon Gamma-1b: Given SC
Period: Overall Study
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2 | Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
Started | 1 | 1 | 1 | 2 | 2
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 2 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Population included all enrolled and treated participants.
Groups:
- Cohort 4 - Cy/Flu + 1 Infusion at DL1 + 1 Infusion at DL2: Following lymphodepleting chemotherapy with fludarabine and cyclophosphamide, patients received FH-MCVA2TCR T-cells at Dose Level 1 IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also received standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells at Dose Level 2.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV Avelumab: Given IV Pembrolizumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2 | Cohort 4 - Cy/Flu + 1 Infusion at DL1 + 1 Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (0) | 63 (0) | 62 (0) | 53 (20) | 70 (4) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 1
  Male | 1 | 1 | 0 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 2 | 2 | 7
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Grade 3 or Higher Determined to be Possibly, Probably or Definitely Secondary to Study Treatments.
Description: Assessed per Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0. Evidence of excessive toxicity will be an observed proportion of toxicities for which the associated lower 80% confidence limit exceeds 40%.
Time Frame: Up to 1 year post infusion
Population: Population included all enrolled and treated participants.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients received FH-MCVA2TCR T-cells at Dose Level 1 IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also received standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells at Dose Level 2.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg
  Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV
  Avelumab: Given IV
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2 | Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
Participants | 0 | 0 | 1 | 2 | 0

2. Primary Outcome: Best Overall Response
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of complete or partial response. Irradiated and non-irradiated lesions will be separately tracked but response determined in totality.
Time Frame: Up to 1 year post infusion
Population: Population included all enrolled and treated participants.
Measure: Number; unit: participants
Groups:
- Cohort 2- Radiation + One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients receive FH-MCVA2TCR T-cells IV at Dose Level 2 over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV Avelumab: Given IV Pembrolizumab: Given IV
- Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients received FH-MCVA2TCR T-cells at Dose Level 1 IV over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also received standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Patients with partial response or stable disease may then receive an additional cycle of FH-MCVA2TCR T-cells at Dose Level 2.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV Avelumab: Given IV Pembrolizumab: Given IV
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2- Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2 | Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0
  Observed Response Rate (CR+PR) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Will be estimated using the method of Kaplan and Meier, with time zero the time of first T cell infusion.
Time Frame: Up to 1 year post infusion
Population: All enrolled and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2: Following treatment with single fraction radiation to a single lesion, patients receive FH-MCVA2TCR T-cells IV at Dose Level 2 over 60-120 minutes. Beginning 14 days after receiving FH-MCVA2TCR T-cells, patients also receive standard of care avelumab IV over 1 hour every 2 weeks for 1 year or pembrolizumab IV over 30 minutes every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  Dose Level 1: 1 x 10^8 FH-MCVATCR T-cells/kg Dose Level 2: Inclusion Range 3.01 x 10^8 - 9.35 x 10^8 FH-MCVATCR T-cells/kg Autologous MCPyV-specific HLA-A02-restricted TCR-transduced CD4+ and CD8+ T-cells FH-MCVA2TCR: Given IV Avelumab: Given IV Pembrolizumab: Given IV
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2 | Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 2
months | 2.8 [NA to NA] — Upper and lower confidence interval for PFS could not be estimated due to insufficient number of events (e.g., participants with disease progression within the time frame for observation). | 0.72 [NA to NA] — Upper and lower confidence interval for PFS could not be estimated due to insufficient number of events (e.g., participants with disease progression within the time frame for observation). | 2.0 [NA to NA] — Upper and lower confidence interval for PFS could not be estimated due to insufficient number of events (e.g., participants with disease progression within the time frame for observation). | 0.92 [0.89 to NA] — Upper confidence interval for PFS could not be estimated due to insufficient number of events (e.g., participants with disease progression within the time frame for observation). | 0.90 [0.82 to NA] — Upper confidence interval for PFS could not be estimated due to insufficient number of events (e.g., participants with disease progression within the time frame for observation).

4. Secondary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan and Meier, with time zero the time of first T cell infusion.
Time Frame: Up to 1 year post infusion
Population: Population included all enrolled and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion at DL1 + One Infusion at DL2 | Cohort 4 - Cy/Flu + One Infusion at DL1 + One Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 2
months | NA [NA to NA] — Due to insufficient number of participants and events (e.g., death), median OS could not be calculated, and upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates. | NA [NA to NA] — Due to insufficient number of participants and events (e.g., death), median OS could not be calculated, and upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates. | 11 [NA to NA] — Due to insufficient number of participants and events (e.g., death), upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates. | 7.6 [6.1 to NA] — Due to insufficient number of participants and events (e.g., death), upper confidence interval for OS could not be obtained using Kaplan-Meier estimates. | NA [NA to NA] — Due to insufficient number of participants and events (e.g., death), median OS could not be calculated, and upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates.

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, serious adverse events, and other (not including serious) adverse events considered related to T Cell infusion were assessed from the time of the first T Cell infusion until the end of study, 12 months total.
Arm/Group | Cohort 1 - Radiation + One Infusion at DL1 | Cohort 2 - Radiation + One Infusion at DL2 | Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2 | Cohort 4 - Cy/Flu + 1 Infusion at DL1 + 1 Infusion at DL2 | Cohort 5 - Interferon Gamma + One Infusion at DL1
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 2/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Radiation + One Infusion at DL1 (N=1) | Cohort 2 - Radiation + One Infusion at DL2 (N=1) | Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2 (N=1) | Cohort 4 - Cy/Flu + 1 Infusion at DL1 + 1 Infusion at DL2 (N=2) | Cohort 5 - Interferon Gamma + One Infusion at DL1 (N=2)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Radiation + One Infusion at DL1 (N=1) | Cohort 2 - Radiation + One Infusion at DL2 (N=1) | Cohort 3 - Radiation + One Infusion DL1 and One Infusion at DL2 (N=1) | Cohort 4 - Cy/Flu + 1 Infusion at DL1 + 1 Infusion at DL2 (N=2) | Cohort 5 - Interferon Gamma + One Infusion at DL1 (N=2)
Altered Mental Status (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White Blood Cell Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03747484/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03747484/ICF_000.pdf